CLINICAL TRIAL: NCT02696525
Title: A Prospective Study of Circulating Tumor DNA Detection in Surveillance for Stage ⅢA Non-small-cell Lung Cancer Patients
Brief Title: Circulating Tumor DNA Detection in Surveillance of Surgical Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: San Valley Biotechnology Incorporated (Unknown)
Responsible Party: Principal Investigator, Jun Wang, Chief，Thoracic Surgery Service, Peking University People's Hospital
Other Study IDs: PTHO1601
Record Dates: First submitted 2016-02-25; First posted 2016-03-02 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Carcinoma; Non-small-cell Lung Cancer; Lung Neoplasms
Keywords: Circulating Tumor DNA; Lung cancer; lead time
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Fresh tumor tissue, urine samples and blood samples were collected from each patient.
  Time:Preoperative, 3 days and 3、6、12、18、24、30、36 months after surgery.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Conduct a prospective study to confirm blood and urine ctDNA detection value in non-small-cell lung cancer patients.

DETAILED DESCRIPTION:
Studies have shown the feasibility of detecting mutation status by blood and urine circulating tumor DNA (ctDNA)in non-small cell lung cancer (NSCLC) patients. However, no prospective has been conducted for usage of ctDNA in postoperative surveillance of NSCLC patients.

We plan to compare tumor makers and radiographic approaches with blood and urine ctDNA in surveillance to assess the lead time of postoperative tumor relapse in stage ⅢA NSCLC patients. And evaluate the correlation between ctDNA level with tumor relapse or metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 80 years
* Undergo radical surgery（R0 resection）
* Histologically confirmed diagnosis of stage ⅢA non-small cell lung cancer
* Positive Driver mutation(EGFR、PTEN、PIK3CA、BRAF、K-RAS、Her2) in tumor tissue
* Blood or urine circulating tumor detect the driver mutation detected in tumor tissue
* Patients must have given written informed consent

Exclusion Criteria:

* Unable to comply with the study procedure
* Malignant tumor history within the past 5 years
* Patients who received any treatment prior to resection
* R1 or R2 resection
* Coexisting small cell lung cancer
* Received target drug therapy after surgery
* Unqualified blood or urine samples

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Histologically confirmed stage ⅢA non-small cell lung cancer patients who have the same driver mutation in tumor tissue and circulating tumor DNA(blood or urine)
Sampling Method: Non-Probability Sample
Enrollment: 145 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Lead time of tumor relapse detection by blood or urine circulation tumor DNA than radiographic approaches | 4 years

SECONDARY OUTCOMES:
Lead time of tumor relapse detection by blood or urine circulation tumor DNA than tumor markers | 4 years
The concordance of ctDNA genomic alterations detection in peripheral blood and urine with those in matched tumor sample | 1 year
Correlation of blood and urine ctDNA concentration before surgery with clinical features and prognosis | 4 years
Correlation of blood and urine ctDNA concentration 3 days after surgery with clinical features and prognosis | 4 years
CtDNA predictive value between locoregional recurrence and distant metastasis | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jun Wang, M.D., Principal Investigator — Peking University People's Hospital; Yilong Wu, M.D., Study Chair — Guang Dong General Hospital; Lin Xu, M.D., Study Director — Jiang Su Cancer Hospital
Locations (3):
- China (3):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Guang Dong General Hospital, Thoracic Surgery, Guangzhou, Guangdong
  - Jiang Su Cancer Hospital, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided